CLINICAL TRIAL: NCT07054021
Title: "Evaluating the Impact of Diverse Antimicrobial Agents on Clinical Outcomes of Various Frenectomy Techniques: A Retrospective Study"
Brief Title: Retrospective Frenectomy Analysis: Techniques and Adjunctive Antimicrobials
Status: Completed | Type: Observational
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, SEVAL CEYLAN ŞEN, asist prof, Saglik Bilimleri Universitesi
Other Study IDs: Seval2
Record Dates: First submitted 2025-06-27; First posted 2025-07-08 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2023-01

CONDITIONS: Frenectomy; Erbium YAG Laser; Antimicrobial Agent
Keywords: frenectomy; erbium yag laser; chlorhexidine; wound healing; visual analog scale

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Conventional Surgery + Postoperative Chlorobene use of mouthwash
- Er:Yag laser surgery + Postoperative use of Chlorobene mouthwash
- Conventional surgery + Postoperative use of Chlorhex plus mouthwash
- Er:Yag laser surgery + Postoperative use of Chlorhex plus mouthwash

SUMMARY:
The frenulum is a mucosal fold that connects the lips and cheeks to the alveolar mucosa or gingiva, with abnormal attachments-particularly papillary and papillary-penetrating types-linked to clinical issues such as gingival recession, diastema, and oral hygiene difficulties. Frenectomy, the complete removal of the frenulum, can be performed using traditional scalpel techniques or soft tissue lasers like Er:YAG, which offers precise cutting with minimal thermal damage. While laser surgery reduces pain and promotes faster healing, it requires careful control and involves higher costs. Postoperative care often includes chlorhexidine-based agents due to their antimicrobial and healing-promoting properties; combinations like Klorhex Plus (chlorhexidine digluconate and flurbiprofen) have demonstrated effectiveness in reducing edema and enhancing wound healing.

DETAILED DESCRIPTION:
The frenulum is a mucosal fold, usually containing closed muscle fibers, that connects the lips and cheeks to the alveolar mucosa and/or gingiva and underlying periosteum. The frenulum problem is most common on the labial surface between the maxillary and mandibular central incisors and in the canine and premolar areas. 1 The labial frenulum restricts and stabilizes lip movement and can also cause gingival recession. 1 Depending on the attachment extension of the fibers, the frenulum is classified as follows: Mucosal; when the frenal fibers are attached up to the mucogingival junction, Gingiva; when fibers are placed inside the attached gingiva, Papillary; when fibers extend towards the interdental papilla, Penetrating the papilla; when the frenal fibers cross the alveolar process and extend to the palatine papilla. 2 Clinically, papillary and papillary-penetrating frenulum are considered pathologic and have been associated with papilla loss, recession, diastema, difficulty in brushing, tooth alignment and psychological disturbances of the individual. 3,4 Frenectomy is the complete removal of the frenulum, including its attachment to the underlying bone. There are two techniques for frenectomy. One is the traditional technique using scalpels and periodontal blades, and the other is the technique using soft tissue lasers. 5,6 Er:YAG is highly effective in cutting soft tissues. Its wavelength is 2940 nm, allowing for shallow penetration and a high water absorption rate. This type of laser can be strongly absorbed by water molecules in the irradiated area, producing a photoelectric effect that causes the water temperature to rise sharply.

Both techniques have some disadvantages; the traditional scalpel technique results in a large rhomboidal wound area at the bottom where primary closure is not possible, and healing occurs with secondary intention. It also causes more pain and discomfort to the patient compared to the laser technique. 7 On the other hand, the laser is an expensive device, and its use requires more precision and control, causing bone necrosis if the beam contacts the bone surface.

Chlorhexidine (CHX) is a cationic bisbiguanide compound with broad-spectrum antimicrobial properties. Although the mouthwash form is most used in dentistry after surgical procedures, gel, spray and dental varnish forms are also preferred for their antiplaque and healing acceleration properties. 8 Klorhex Plus mouthwash, containing 0.5 g flurbiprofen and 0.24 g chlorhexidine digluconate has also been shown to have significant contributions in reducing edema and accelerating wound healing in oral wounds.9

ELIGIBILITY:
Inclusion Criteria:

* Patients who presented to the Department of Periodontology, Gülhane Faculty of Dentistry between January 1, 2023, and March 1, 2025, and underwent maxillary labial frenectomy.
* Patients from whom a complete and signed surgical informed consent form was obtained.
* Patients with complete clinical measurements recorded at baseline, and on postoperative days 7, 14, and 28.
* Patients whose wound healing was scored using the Landry Wound Healing Index and documented on days 7, 14, and 28 postoperatively.
* Patients whose epithelialization status was evaluated and documented on postoperative days 7, 14, and 28.
* Patients who received one of the following treatment protocols:
* Conventional surgery + postoperative use of Kloroben mouthwash,
* Er:YAG laser surgery + postoperative use of Kloroben mouthwash,
* Conventional surgery + postoperative use of Klorhex Plus mouthwash,
* Er:YAG laser surgery + postoperative use of Klorhex Plus mouthwash.
* Patients who completed a written pain assessment using the Visual Analog Scale (VAS) daily for one week postoperatively.
* Patients who documented postoperative bleeding and the number of analgesic intakes in written form.

Exclusion Criteria:

* Patients who presented to the Department of Periodontology, Gülhane Faculty of Dentistry between January 1, 2023, and March 1, 2025, and underwent mandibular labial frenectomy.
* Patients with incomplete or missing surgical informed consent forms.
* Patients for whom clinical measurements, Landry wound healing scores, and hydrogen peroxide (H₂O₂) tests were not performed.
* Patients treated with diode laser.
* Patients whose postoperative VAS pain records, number of analgesics used, and bleeding status were not documented.
* Patients who received postoperative antibiotic therapy.
* Patients who did not use Kloroben or Klorhex Plus mouthwash postoperatively.

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Among 463 patients who applied to Gülhane Faculty of Dentistry, Department of Periodontology for frenectomy indication between January 2023 and March 2025, a total of 102 patients who were treated with the traditional method and Er:Yag laser were included in the study.
Sampling Method: Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2025-05-15 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2025-05-15 (Actual)

PRIMARY OUTCOMES:
Wound healing (WHI) was used as the primary outcome measure. | The WHI was recorded on the 7th, 14th and 28th days.
  Wound healing was scored according to WHI 14. The WHI was recorded on the 7th, 14th and 28th days. The primary outcome of the study was to measure the palatal wound healing status using the WHI, which grades the wound healing on a scale. This index, which has a score range of 1 (very poor) to 5 (excellent), evaluates tissue color, response to palpation, granulation tissue presence, incision margins' epithelialization, and amount of suppuration

SECONDARY OUTCOMES:
Postoperative pain was evaluated as a secondary outcome. | The secondary results of the study showed that patients' perceptions of pain after surgical procedures were rated on a numerical rating scale from; VAS 0 (no pain) and 100 (the most severe pain imaginable) between days 1 and 7 and post-surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Health Sciences University Gulhane Faculty of Dentistry, Ankara, KEÇİÖREN, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
It will not be shared as it contains personal data belonging to patients.